CLINICAL TRIAL: NCT04576000
Title: PhaRmacOkinetics and PHarmacodynamic BiomarkErs of Janus Kinase Inhibitor Therapy in PatIents With Ulcerative Colitis (PROPHETIC)
Brief Title: Identification of Biomarkers of Janus Kinase Inhibitor Therapy in Patients With Ulcerative Colitis
Acronym: PROPHETIC
Status: Terminated | Type: Observational
Why Stopped: Not able to meet recruitment targets
Sponsor: Alimentiv Inc. (Other)
Collaborators: Alimentiv Translational Research Consortium (Unknown)
Responsible Party: Sponsor
Other Study IDs: RP1907
Record Dates: First submitted 2020-09-17; First posted 2020-10-05 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Janus Kinase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, fecal, and colonic tissue sampling
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Open-Label Group: Eligible patients will include those who will be prescribed Janus Kinase inhibitor as part of their routine medical care.
  Interventions: Drug: Janus Kinase Inhibitor

INTERVENTIONS:
Drug: Janus Kinase Inhibitor — Janus Kinase inhibitor induction therapy will be administered according to Standard Of Care (SOC)

SUMMARY:
This study aims to provide new mechanistic insights into the molecular determinants of response or nonresponse to Janus Kinase inhibitor therapy and the biological heterogeneity that exists in Ulcerative Colitis. This study will include patients who are initiating Janus Kinase inhibitor therapy according to standard of care. This study consists of:

* Part 1: 8 or 10 week induction therapy followed by an 8-week maintenance therapy
* Part 2: Patients who continue Janus Kinas inhibitor therapy after part 1 will be followed further for a total of 2 years, or until discontinuation of Janus Kinase inhibitor therapy (whichever is first)

ELIGIBILITY:
Inclusion Criteria:

1.18 years of age or older.

2.Male or nonpregnant, nonlactating females.

3.Diagnosis of Ulcerative Colitis for at least 3 months prior to screening.

4.Moderately to severely active Ulcerative Colitis (total Mayo Clinic Score ≥ 6), with objective evidence of inflammation defined by a Mayo endoscopic subscore (MES) ≥ 2 and disease extending > 15 cm from the anal verge.

5.Physician plans to administer Janus Kinase inhibitor for at least 8 weeks of induction therapy as part of Standard of Care (SOC).

6.Documentation of a negative test result for latent tuberculosis within the last 12 months, or according to routine clinical practice.

7.Able to participate fully in all aspects of this clinical trial, including collection of tissue biopsies.

8.Written informed consent must be obtained and documented.

Exclusion Criteria:

1. Diagnosis of Crohn's disease or indeterminate colitis.
2. An active, serious infection, including localized infections.
3. Concomitant administration of biological therapies for Ulcerative Colitis or potent immunosuppressants, such as azathioprine and cyclosporine. Subjects with previous exposure to these treatments should undergo an appropriate washout period according to local practice prior to starting Janus Kinase inhibitor, in keeping with routine clinical practice.
4. Hematology laboratory (e.g., absolute lymphocyte count, absolute neutrophil count, and hemoglobin that contraindicate the product label.
5. Interval between live vaccinations and initiation of tofacitinib therapy should be in accordance with current vaccination guidelines regarding immunosuppressive agents.
6. Serious underlying disease other than Ulcerative Colitis that in the opinion of the investigator may interfere with the subject's ability to participate fully in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve subjects with moderately to severely active Ulcerative Colitis who will receive Janus Kinase inhibitor for at least 8 weeks, followed by Janus Kinase inhibitor maintenance therapy for an additional 8 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Identify predictive fecal biomarkers that are associated with a change from baseline in UC-100 score | 8 or 10 weeks; 24 weeks
  The UC-100 is a composite disease activity index consisting of clinical, endoscopic, and histological findings. The UC-100 is calculated by summing the weighted Mayo Clinic Score (MCS) stool frequency and endoscopy subscores, and the Robarts Histopathology Index (RHI) score as follows: UC-100 Score = 1 + (16 X stool frequency) + (6 X endoscopic subscore) + (RHI score). The total UC-100 score ranges from 1 to 100, with higher scores representing more severe disease activity.
Identify predictive blood biomarkers that are associated with a change from baseline in UC-100 score | 8 or 10 weeks; 24 weeks
Identify predictive tissue biomarkers that are associated with a change from baseline in UC-100 score | 8 or 10 weeks; 24 weeks

SECONDARY OUTCOMES:
Identify pharmacodynamic fecal biomarkers that are associated with a change from baseline in UC-100 score | 8 or 10 weeks, 24 weeks
Identify pharmacodynamic blood biomarkers that are associated with a change from baseline in UC-100 score | 8 or 10 weeks, 24 weeks
Identify pharmacodynamic tissue biomarkers that are associated with a change from baseline in UC-100 score | 8 or 10 weeks, 24 weeks
Identify a fecal biomarker signature as a surrogate measure for change from baseline in UC-100 score | 8 or 10 weeks, 24 weeks
Identify a blood biomarker signature as a surrogate measure for change from baseline in UC-100 score | 8 or 10 weeks, 24 weeks
Identify a tissue biomarker signature as a surrogate measure for change from baseline in UC-100 score | 8 or 10 weeks, 24 weeks
Identify whether colonic tissue pSTAT at week 8 and/or 24 correlates with change from baseline in UC-100 score | 8 or 10 weeks, 24 weeks
Determine the time-concentration profile of Janus Kinase inhibitor at steady state in stool samples. | 24 weeks
Determine the time-concentration profile of Janus Kinase inhibitor at steady state in serum samples. | 24 weeks
Determine the time-concentration profile of Janus Kinase inhibitor at steady state in tissue samples. | 24 weeks
Evaluate correlation of exposure of Janus Kinase inhibitor between stool samples following SOC induction therapy and at Week 24. | 8 or 10 weeks, 24 weeks
Evaluate correlation of exposure of Janus Kinase inhibitor between serum samples following SOC induction therapy and at Week 24. | 8 or 10 weeks, 24 weeks
Evaluate correlation of exposure of Janus Kinase inhibitors between tissue samples following SOC induction therapy and at Week 24. | 8 or 10 weeks, 24 weeks
Explore the exposure-response relationship of Janus Kinase inhibitors with exposure measured in stool samples and response defined as tissue PD biomarkers following SOC induction therapy and at Week 24. | 8 or 10 weeks, 24 weeks
Explore the exposure-response relationship of Janus Kinase inhibitors with exposure measured in serum samples and response defined as tissue PD biomarkers following SOC induction therapy and at Week 24. | 8 or 10 weeks, 24 weeks
Explore the exposure-response relationship of Janus Kinase inhibitors with exposure measured in tissue samples and response defined as tissue PD biomarkers following SOC induction therapy and at Week 24. | 8 or 10 weeks, 24 weeks
Develop an exposure-response model of Janus Kinase inhibitors to characterize the relationships between local and systemic drug exposure and clinical, endoscopic, histologic, or biologic response to therapy. | 24 weeks
Identify potential demographic and disease factors affecting the most relevant JAKi exposure-response relationships and determine target threshold of systemic exposure associated with relevant clinical, endoscopic, histologic, and/or biologic outcomes. | 8 or 10 weeks, 24 weeks
Evaluate long-term hospitalization rates, surgery rates, and corticosteroid use after initiation of Janus Kinase inhibitor therapy and identify baseline or early biomarker signatures associated with these long-term healthcare resource use outcomes | 2 years
Measure adverse drug reactions, clinical, endoscopic, and histologic response and remission rates to Janus Kinase inhibitors in a "real-world" population | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vipul Jairath, MD, PhD, Principal Investigator — Alimentiv Inc.
Locations (1):
- Amsterdam Medical Center, IBD Center, Amsterdam, North Halland, Netherlands

REFERENCES:
- [Background] Jairath V, Jeyarajah J, Zou G, Parker CE, Olson A, Khanna R, D'Haens GR, Sandborn WJ, Feagan BG. A composite disease activity index for early drug development in ulcerative colitis: development and validation of the UC-100 score. Lancet Gastroenterol Hepatol. 2019 Jan;4(1):63-70. doi: 10.1016/S2468-1253(18)30306-6. Epub 2018 Oct 18. PMID 30343116
- [Background] Mosli MH, Feagan BG, Zou G, Sandborn WJ, D'Haens G, Khanna R, Shackelton LM, Walker CW, Nelson S, Vandervoort MK, Frisbie V, Samaan MA, Jairath V, Driman DK, Geboes K, Valasek MA, Pai RK, Lauwers GY, Riddell R, Stitt LW, Levesque BG. Development and validation of a histological index for UC. Gut. 2017 Jan;66(1):50-58. doi: 10.1136/gutjnl-2015-310393. Epub 2015 Oct 16. PMID 26475633
- [Background] Scherl EJ, Pruitt R, Gordon GL, Lamet M, Shaw A, Huang S, Mareya S, Forbes WP. Safety and efficacy of a new 3.3 g b.i.d. tablet formulation in patients with mild-to-moderately-active ulcerative colitis: a multicenter, randomized, double-blind, placebo-controlled study. Am J Gastroenterol. 2009 Jun;104(6):1452-9. doi: 10.1038/ajg.2009.83. Epub 2009 Apr 21. PMID 19491859
- [Background] Salas A, Hernandez-Rocha C, Duijvestein M, Faubion W, McGovern D, Vermeire S, Vetrano S, Vande Casteele N. JAK-STAT pathway targeting for the treatment of inflammatory bowel disease. Nat Rev Gastroenterol Hepatol. 2020 Jun;17(6):323-337. doi: 10.1038/s41575-020-0273-0. Epub 2020 Mar 19. PMID 32203403